CLINICAL TRIAL: NCT01539512
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Idelalisib (GS-1101) in Combination With Rituximab for Previously Treated Chronic Lymphocytic Leukemia
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Study of Idelalisib in Combination With Rituximab for Previously Treated Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-312-0116; 2011-005180-24 (EudraCT Number)
Record Dates: First submitted 2012-02-12; First posted 2012-02-27 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2015-04

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; CAL-101; GS 1101; PI3K; GS-US-312-0117; idelalisib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — idelalisib; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Idelalisib + rituximab (Active Comparator): Participants will receive idelalisib plus rituximab
  Interventions: Drug: Idelalisib; Drug: Rituximab
- Placebo + rituximab (Placebo Comparator): Participants will receive placebo to match idelalisib plus rituximab
  Interventions: Drug: Rituximab; Drug: Placebo to match idelalisib

INTERVENTIONS:
Drug: Idelalisib — Idelalisib 150 mg tablet administered orally twice daily
  Other Names: Zydelig®; GS-1101; CAL 101
  Arms: Idelalisib + rituximab
Drug: Rituximab — Rituximab administered intravenously 8 times through Week 20: Day 1: 375 mg/m^2, and 500 mg/m^2 thereafter
  Other Names: Rituxan®
Drug: Placebo to match idelalisib — Placebo to match idelalisib administered orally twice daily
  Arms: Placebo + rituximab

SUMMARY:
This Phase 3, randomized, double-blind, placebo-controlled study is to evaluate the effect of idelalisib in combination with rituximab on the onset, magnitude, and duration of tumor control in participants previously treated for chronic lymphocytic leukemia (CLL). Eligible patients will be randomized with a 1:1 ratio into 1 of the 2 treatment arms to receive either idelalisib plus rituximab or placebo plus rituximab. Participants who are tolerating primary study therapy but experience definitive CLL progression are eligible to receive active idelalisib therapy in the extension study, GS-US-312-0117.

ELIGIBILITY:
Inclusion:

* Adult subjects with previously treated recurrent CLL who have measurable lymphadenopathy
* Require therapy for CLL
* Have experienced CLL progression < 24 months since the completion of the last prior therapy
* Currently not sufficiently fit to receive cytotoxic therapy because of chemotherapy-induced bone marrow damage or comorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jahn, MD, Study Director — Gilead Sciences
Locations (72):
- United States (34):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Arizona Oncology Associates, Tucson, Arizona
  - University of California, San Diego- Moores Cancer Center, La Jolla, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - UCLA, Santa Monica, California
  - Stanford Cancer Center, Stanford, California
  - Rocky Mountain Blood and Marrow Transplant Program, Denver, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Collaborative Medical Research Corporation, Boynton Beach, Florida
  - Collaborative Research Group LLC, Boynton Beach, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - University of Florida, Gainesville, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Hematology Oncology Associates of Northern New Jersey, Morristown, New Jersey
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Willamette Valley Cancer Center, Springfield, Oregon
  - Northwest Cancer Specialists, PC, Tualatin, Oregon
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Texas Oncology, P.A., Fort Worth, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - Cancer Care Network of South Texas, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc, Roanoke, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Yakima Valley Memorial Hospital / North Star Lodge, Yakima, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (7):
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Régional Universitaire de Lille (CHRU), Lille
  - Hôpital Emile Muller, Mulhouse
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Hopital Purpan, Toulouse
- Germany (6):
  - Universitätsklinikum Köln, Cologne
  - Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Internistische Gemeinschaftspraxis, Erlangen
  - Stauferklinikum Schwäb. Gmünd, Mutlangen
  - Hämatologische/Onkologische Gemeinschaftspraxis Dr. Peter Schmidt / Dr. Holger Klaproth, Neunkirchen
  - Universitätsklinikum Ulm, Ulm
- Italy (3):
  - Ospedale Oncologico Regionale A. Businco, Cagliari
  - Ospedale San Raffaele S.r.l., Milan
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- United Kingdom (22):
  - Royal Bournemouth Hospital, Bournemouth
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Castle Hill Hospital, Cottingham
  - Dorset County Hospital, Dorchester
  - Western General Hospital, Edinburgh
  - Northwick Park Hospital, Harrow
  - St James's University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - King's College Hospital, London
  - Hammersmith Hospital, London
  - Sarah Cannon Research Institute UK, London
  - Freeman Hospital, Newcastle upon Tyne
  - Princess Royal University Hospital, Orpington
  - Salisbury District Hospital, Salisbury
  - Southampton General Hospital, Southampton
  - Royal Marsden Hospital, Sutton
  - Great Western Hospital, Swindon
  - Torbay District General Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - New Cross Hospital, Wolverhampton
  - Yeovil District Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Barrientos JC, Hillmen P, Salles G, Sharman J, Stilgenbauer S, Gurtovaya O, Xing G, Ruzicka B, Bhargava P, Ghia P, Pagel JM. No increased bleeding events in patients with relapsed chronic lymphocytic leukemia and indolent non-Hodgkin lymphoma treated with idelalisib. Leuk Lymphoma. 2021 Apr;62(4):837-845. doi: 10.1080/10428194.2020.1845339. Epub 2020 Dec 10. PMID 33297794
- [Derived] Gordon MJ, Huang J, Chan RJ, Bhargava P, Danilov AV. Medical comorbidities in patients with chronic lymphocytic leukaemia treated with idelalisib: analysis of two large randomised clinical trials. Br J Haematol. 2021 Feb;192(4):720-728. doi: 10.1111/bjh.16879. Epub 2020 Jun 29. PMID 32599655
- [Derived] Furman RR, Sharman JP, Coutre SE, Cheson BD, Pagel JM, Hillmen P, Barrientos JC, Zelenetz AD, Kipps TJ, Flinn I, Ghia P, Eradat H, Ervin T, Lamanna N, Coiffier B, Pettitt AR, Ma S, Stilgenbauer S, Cramer P, Aiello M, Johnson DM, Miller LL, Li D, Jahn TM, Dansey RD, Hallek M, O'Brien SM. Idelalisib and rituximab in relapsed chronic lymphocytic leukemia. N Engl J Med. 2014 Mar 13;370(11):997-1007. doi: 10.1056/NEJMoa1315226. Epub 2014 Jan 22. PMID 24450857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 53 study sites in the United States and Europe. The first participant was screened on 03 April 2012. The last study visit occurred on 20 April 2014.
Groups:
- Idelalisib + Rituximab: Idelalisib 150 mg tablet administered orally twice daily plus rituximab (8 intravenous doses through Week 20: Day 1: 375 mg/m^2, and 500 mg/m^2 thereafter)
- Placebo + Rituximab: Placebo to match idelalisib administered orally twice daily plus rituximab (8 intravenous doses through Week 20: Day 1: 375 mg/m^2, and 500 mg/m^2 thereafter)
Period: Overall Study
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Started | 110 | 110
Completed | 87 (Completed=reached primary efficacy endpoint (progressive disease or death) or finished study period.) | 97 (Completed=reached primary efficacy endpoint (progressive disease or death) or finished study period.)
Not Completed | 23 | 13
Not completed — Adverse Event | 9 | 7
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 12 | 5
Not completed — Richter's Transformation | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Analysis Set: randomized participants with treatment group designated according to initial randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab | Total
Number analyzed (Participants) | 110 | 110 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (7.7) | 70 (8.1) | 71 (7.9)
Age, Customized [Number; unit: participants]
  < 65 years | 21 | 27 | 48
  ≥ 65 years | 89 | 83 | 172
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 42 | 76
  Male | 76 | 68 | 144
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 101 | 102 | 203
  Not Permitted | 6 | 6 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  White | 100 | 98 | 198
  Black or African American | 3 | 3 | 6
  Other | 2 | 2 | 4
  Not Permitted | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  France | 3 | 3 | 6
  Germany | 7 | 5 | 12
  Italy | 2 | 5 | 7
  United Kingdom | 18 | 14 | 32
  United States | 80 | 83 | 163
Karnofsky Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0-100; the lower the score, the worse the survival for most serious illnesses.
  participants
    40 | 1 | 1 | 2
    50 | 3 | 4 | 7
    60 | 6 | 5 | 11
    70 | 20 | 13 | 33
    80 | 42 | 46 | 88
    90 | 23 | 28 | 51
    100 | 15 | 13 | 28
Time Since Diagnosis [Mean (Standard Deviation); unit: months] | 108.3 (62.28) | 106.4 (52.73) | 107.4 (57.58)
Rai Stage at Screening [Number; unit: participants] — Rai staging categorizes the disease progression of chronic lymphocytic leukemia (CLL), with classifications of low- (Stage 0), intermediate- (Stage 1 and 2), and high-risk (Stages 3 and 4) categories. Rai Stage 0: high number of lymphocytes in the blood (lymphocytosis) only. Rai Stage 1: lymphocytosis with enlarged lymphoid tissues (lymphadenopathy). Rai Stage 2: lymphocytosis with enlarged liver (hepatomegaly) or spleen (splenomegaly). Rai Stage 3: lymphocytosis with low red blood cell count (anemia). Rai Stage 4: lymphocytosis with low number of blood platelets (thrombocytopenia).
  participants
    Rai Stage 0 | 0 | 1 | 1
    Rai Stage 1 | 18 | 19 | 37
    Rai Stage 2 | 16 | 10 | 26
    Rai Stage 3 | 22 | 18 | 40
    Rai Stage 4 | 48 | 54 | 102
    Missing | 6 | 8 | 14
Binet Stage at Screening [Number; unit: participants] — Binet staging classifies CLL according to the number of lymphoid tissues involved, as well as the presence of anemia or thrombocytopenia. Stage A: fewer than three areas of enlarged lymphoid tissue; enlarged lymph nodes of the neck, underarms, and groin, as well as the spleen, are each considered "one group" whether unilateral (one-sided) or bilateral (on both sides). Binet Stage B: more than three areas of enlarged lymphoid tissue. Binet Stage C: anemia plus thrombocytopenia.
  participants
    Binet Stage A | 7 | 4 | 11
    Binet Stage B | 29 | 32 | 61
    Binet Stage C | 63 | 60 | 123
    Missing | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression-free survival was defined as the interval from randomization to the earlier of the first documentation of definitive disease progression or death from any cause. Definitive disease progression was CLL progression based on standard criteria (other than lymphocytosis alone) as defined by the 2008 update of the International Workshop on CLL guidelines, ie, appearance of any new lesion; increase by ≥ 50% in the sum of the products of the perpendicular diameters of measured lymph nodes (SPD); new or ≥ 50% enlargement of liver or spleen; transformation to a more aggressive histology (eg, Richter's or prolymphocytic transformation); reduction in the number of blood cells (cytopenia) attributable to CLL.
Time Frame: Up to 17 months
Population: Intent-to-Treat (ITT) Analysis Set: randomized participants with treatment group designated according to initial randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 110 | 110
months | NA [10.7 to NA] — NA = Not reached due to insufficient number of events | 5.5 [3.8 to 7.1]
Statistical Analysis 1: Comparison: Idelalisib + Rituximab vs Placebo + Rituximab; Test type: Superiority or Other; p < 0.0001, Log Rank; P-value is from stratified log-rank test, adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.18, 95% CI 2-sided [0.10 to 0.32]

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate was defined as the percentage of participants who achieved a best overall response of complete response or partial response.
  Complete response was defined as no lymphadenopathy, hepatomegaly, splenomegaly; normal complete blood count; confirmed by bone marrow aspirate & biopsy.
  Partial response was defined as >1 of the following criteria: a 50% decrease in peripheral blood lymphocytes, lymphadenopathy, liver size, spleen size; plus ≥ 1 of the following: ≥ 1500/μL absolute neutrophil count, > 100000/μL platelets, > 11.0 g/dL hemoglobin or 50% improvement for either of these parameters without transfusions or growth factors.
Time Frame: Up to 17 months
Population: ITT Analysis Set: randomized participants with treatment group designated according to initial randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 110 | 110
percentage of participants | 74.5 [65.4 to 82.4] | 14.5 [8.5 to 22.5]

3. Secondary Outcome: Lymph Node Response Rate
Description: Lymph node response rate was defined as the percentage of participants who achieved a ≥ 50% decrease from baseline in the SPD of index lymph nodes.
Time Frame: Up to 17 months
Population: ITT Analysis Set: randomized participants with treatment group designated according to initial randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 110 | 110
percentage of participants | 92.2 [85.1 to 96.6] | 5.9 [2.2 to 12.5]

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval from randomization to death from any cause.
Time Frame: Up to 17 months
Population: ITT Analysis Set: randomized participants with treatment group designated according to initial randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 110 | 110
months | NA [NA to NA] — NA = Not reached due to insufficient number of events | NA [12.8 to NA] — NA = Not reached due to insufficient number of events
Statistical Analysis 1: Comparison: Idelalisib + Rituximab vs Placebo + Rituximab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.28, 95% CI 2-sided [0.11 to 0.69]

5. Secondary Outcome: Complete Response Rate
Description: Complete response rate was defined as the percentage of participants who achieved a complete response.
Time Frame: Up to 17 months
Population: ITT Analysis Set: randomized participants with treatment group designated according to initial randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 110 | 110
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: During study treatment plus 30 days (up to 2 years)
Description: Safety Analysis Set: randomized participants who received at least 1 dose of study drug, with treatment assignments designated according to the actual treatment received.
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Serious Adverse Events (participants affected / at risk) | 65/110 | 43/108
Other Adverse Events (participants affected / at risk) | 103/110 | 102/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Rituximab (N=110) | Placebo + Rituximab (N=108)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 6
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 0
Gastric mucosa erythema (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 3
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Device dislocation (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 2
Pyrexia (General disorders) | 10 | 3
Abscess limb (Infections and infestations) | 0 | 1
Alpha haemolytic streptococcal infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 4
Diverticulitis (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Fungal oesophagitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster disseminated (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Listeriosis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Lung infection (Infections and infestations) | 3 | 1
Mucosal infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 13 | 10
Pneumonia fungal (Infections and infestations) | 2 | 0
Pneumonia legionella (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 7 | 3
Sepsis syndrome (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 0 | 2
Soft tissue infection (Infections and infestations) | 0 | 1
Stenotrophomonas infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2
Blood creatinine increased (Investigations) | 0 | 2
International normalised ratio increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Iiird nerve disorder (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Rituximab (N=110) | Placebo + Rituximab (N=108)
Anaemia (Blood and lymphatic system disorders) | 13 | 11
Neutropenia (Blood and lymphatic system disorders) | 28 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 9 | 11
Abdominal pain upper (Gastrointestinal disorders) | 8 | 3
Colitis (Gastrointestinal disorders) | 6 | 1
Constipation (Gastrointestinal disorders) | 16 | 15
Diarrhoea (Gastrointestinal disorders) | 31 | 19
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 0
Nausea (Gastrointestinal disorders) | 30 | 25
Stomatitis (Gastrointestinal disorders) | 7 | 1
Vomiting (Gastrointestinal disorders) | 16 | 9
Asthenia (General disorders) | 8 | 8
Chills (General disorders) | 27 | 16
Fatigue (General disorders) | 34 | 35
Oedema peripheral (General disorders) | 12 | 10
Pain (General disorders) | 8 | 1
Pyrexia (General disorders) | 40 | 18
Bronchitis (Infections and infestations) | 7 | 4
Cellulitis (Infections and infestations) | 7 | 2
Pneumonia (Infections and infestations) | 4 | 6
Sinusitis (Infections and infestations) | 9 | 6
Upper respiratory tract infection (Infections and infestations) | 9 | 13
Urinary tract infection (Infections and infestations) | 8 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 21 | 33
Alanine aminotransferase increased (Investigations) | 8 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 0
Weight decreased (Investigations) | 11 | 9
Decreased appetite (Metabolism and nutrition disorders) | 18 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 7
Dizziness (Nervous system disorders) | 7 | 9
Headache (Nervous system disorders) | 11 | 9
Anxiety (Psychiatric disorders) | 3 | 7
Insomnia (Psychiatric disorders) | 10 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 22
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 12 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 5
Rash (Skin and subcutaneous tissue disorders) | 16 | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 7
Hypotension (Vascular disorders) | 4 | 7

LIMITATIONS AND CAVEATS:
Following a recommendation by an independent Data Monitoring Committee (DMC), the study was stopped early due to highly statistically significant results for the primary efficacy endpoint of progression-free survival.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years